CLINICAL TRIAL: NCT05843149
Title: Manual Therapy/Exercises vs. Physiotherapy/Back School vs. Waiting List in Patients With Chronic Low Back Pain - a Randomized Controlled Trial
Brief Title: Manual Therapy/Exercises vs. Physiotherapy/Back School vs. Waiting List in Patients With Chronic Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor did not want to continue the study.
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHKManual
Record Dates: First submitted 2023-04-20; First posted 2023-05-06 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual Therapy/Exercises (Experimental): Three individual therapy sessions and nine group sessions manual therapy/exercises of 60 min. duration under the guidance of a trained therapist.
  Interventions: Behavioral: Manual Therapy/Exercises
- Physiotherapy/Back School (Experimental): Three individual therapy sessions and nine group sessions physiotherapy/back school of 60 min. duration under the guidance of a trained therapist.
  Interventions: Behavioral: Physiotherapy/Back School
- Waiting List (No Intervention): Study arm 3 consists of a waiting list control group, combined with the offer to participate in one of the above mentioned interventions after 6 months.

INTERVENTIONS:
Behavioral: Manual Therapy/Exercises — Three individual therapy sessions and nine group sessions manual therapy/exercises of 60 min. duration under the guidance of a trained therapist.
  Arms: Manual Therapy/Exercises
Behavioral: Physiotherapy/Back School — Three individual therapy sessions and nine group sessions physiotherapy/back school of 60 min. duration under the guidance of a trained therapist.
  Arms: Physiotherapy/Back School

SUMMARY:
A randomized controlled trial for patients with chronic low back pain with two treatment arms and one waiting list control group. Primary outcome is pain intensity on VAS.

ELIGIBILITY:
Inclusion Criteria:

* pre-existing and specialist confirmed diagnosis of chronic low back pain for at least 3 months prior to inclusion
* Average pain intensity with at least 40 mm on the VAS from 0 to 100 mm and pain on at least 5 of 7 weekdays in the last 3 months.

Exclusion criteria:

* Regular own exercise practice for the treatment of back pain (including yoga and other interventions)
* Invasive spinal procedures within the past 6 weeks or planned within the next 10 weeks
* Acute disc herniation (diagnosed within the last 3 months)
* Congenital deformities of the lumbar spine
* Rheumatoid arthritis
* Fibromyalgia
* Ankylosing spondylitis
* Severe comorbidities
* Pregnancy/lactation
* Current participation in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average pain intensity in previous week | 3 months
  Intensity of pain in previous week as measured on a 100 mm visual analog scale (0-100).

SECONDARY OUTCOMES:
Change from baseline for back pain specific disability | 3 months, 6 months
  Use of standardized Roland Morris Disability Questionnaire (RMDQ) to assess back pain specific disability. The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline in average pain intensity in previous week | 6 months
  Intensity of pain in previous week as measured on a 100 mm visual analog scale (0-100).
Change from baseline in pain bothersomeness in previous week | 3 months, 6 months
  Bothersomeness in previous week as measured on a 100 mm visual analog scale (0-100).
Change from baseline in pain medication use in the previous week | 3 months, 6 months
  Specific self-reported pain medication use in previous week.
Change from baseline for health related quality of life | 3 months, 6 months
  Use of standardized Short Form 36 Health Survey (SF-36). The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline for pain self-efficacy | 3 months, 6 months
  Use of standardized Pain Self-Efficacy Questionnaire (PSEQ). The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline for work productivity | 3 months, 6 months
  Use standardized Work Productivity and Activity Impairment Questionnaire (WPAI) to assess employment status and productivity. The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Change from baseline for anxiety and depression | 3 months, 6 months
  Use of standardized Hospital Anxiety and Depression Scale (HADS). The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.

OTHER OUTCOMES:
Number of participants with adverse events as a measure of safety and treatment adherence | 3 months, 6 months
  Identify and assess self reported and unanticipated adverse events over the course of the study as a measure of safety and treatment adherence.
Treatment adherence (class/session attendance) | 3 months, 6 months
  Assess treatment adherence according to attendance during 12 week intervention period.
App via mobile phones | 3 times daily within baseline and 6 months
  Use of an mobile app to assess back pain intensity, pain medication, practice time

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided